CLINICAL TRIAL: NCT06885151
Title: A New Website for Australian IVF Patients 'Evidence-based IVF': an Online Randomised Trial
Brief Title: A New Website for Australian IVF Patients: 'Evidence-based IVF'
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Responsible Party: Principal Investigator, Sarah Lensen, Senior Research Fellow, Principal Investigator, University of Melbourne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2025-31333
Record Dates: First submitted 2025-03-05; First posted 2025-03-20 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-03

CONDITIONS: IVF; IVF Treatment; IVF-ET; IVF/ICSI
Keywords: IVF add-ons; Evidence-based IVF

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Evidence-based IVF information (Experimental): Evidence-based IVF information
  Interventions: Other: Evidence-based IVF website content
- Control (Active Comparator): Control information
  Interventions: Other: Control

INTERVENTIONS:
Other: Evidence-based IVF website content — The Evidence-based IVF website has been developed through a robust co-design process with IVF patients and clinicians, and the information about effectiveness and safety of add-ons was produced following established systematic review methodology of Cochrane (including risk of bias, GRADE, and TRACT assessment). They will view information about one of the following IVF add-ons: Endometrial receptivity array (ERA test), EmbryoGlue, or intralipid.
  Arms: Evidence-based IVF information
Other: Control — Participants will view information that has been generated by combining information from the top 3 websites retrieved on Google search of the add-on name. They will view information about one of the following IVF add-ons: Endometrial receptivity array (ERA test), EmbryoGlue, or intralipid.
  Arms: Control

SUMMARY:
IVF 'add-ons' are extra procedures, techniques, or medicines offered alongside standard IVF treatments, often marketed to improve success rates. Examples include EmbryoGlue, endometrial scratching, and acupuncture. However, most lack clear evidence of effectiveness or safety. Despite this, over 80% of Australian IVF patients use add-ons, sometimes paying thousands of dollars.

Patients often rely on clinic websites and online forums for information, but these sources frequently exaggerate benefits while omitting information about costs and risks. There is no independent, evidence-based resource in Australia to guide decision-making, a gap recognized by both patients and government reports.

To address this, the investigators developed "Evidence-Based IVF (EBI)," a new website informed by patient decision aid standards, expertise in digital health and risk communication, and co-design sessions with IVF patients and professionals. The investigators now plan to evaluate how well it helps patients understand the evidence base for IVF add-ons.

DETAILED DESCRIPTION:
In response to widespread calls for evidence-based resources about IVF options and add-ons in Australia, the investigators assembled a multidisciplinary team to co-design a novel website prototype referred to as 'Evidence-based IVF (EBI)'. Informed by patient decision aids standards, the MAGIC App, and applying the investigators' expertise in digital and risk communication and evidence-informed health decisions, the investigators undertook interviews with Australian IVF patients and professionals to test and iteratively modify a new resource. This trial will evaluate how this website performs in terms of gist knowledge and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Live in Australia
* Undergone IVF/embryo transfer in the last 2 years or planning IVF/embryo transfer in the next six months. IVF refers to any IVF/ICSI/embryo transfer cycle in which the participant or their partner is planning to get pregnant.

Exclusion Criteria:

* People who underwent IVF process for egg-freezing or embryo freezing and not intending to conceive, or who received an embryo transfer as a surrogate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1217 (Actual)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-04-06 (Actual); Study Completion 2025-04-06 (Actual)

PRIMARY OUTCOMES:
Gist comprehension using bespoke 5-item questionnaire | 24 hours
  5-item measure, correct answer = 2 points per item, max of 10 points, higher score means better comprehension
  Items 1-3. How does [EmbryoGlue/Intralipid/ERA test] affect the chance of [getting pregnant/having a baby/having a miscarriage] from IVF?
  * Increases the chance
  * Possibly increases the chance
  * Has no effect on the chance
  * Possibly decreases the chance
  * Decreases the chance
  * Its unclear
  * I don't know
    4. The scientific studies of [EmbryoGlue/Intralipid/ERA test] are
  * High quality and very reliable
  * Moderate quality and reliable
  * Low quality and somewhat reliable
  * Very low quality and not at all reliable
  * I don't know
    5. [EmbryoGlue/Intralipid/ERA test] is associated with the following risks
  * Headache
  * Infection
  * Pain or discomfort
  * Nausea and vomiting
  * Fever or chills
  * Hair loss
  Developed from Smith 2012

SECONDARY OUTCOMES:
Proportion of participants with correct comprehension of magnitude of effect | 24 hours
  An assessment of understanding of the magnitude of possible benefit as an absolute risk difference.
  "For every 100 people having IVF, roughly how many more would [get pregnant/have a baby/have a miscarriage] using EmbryoGlue?
  * 5 more
  * 10 more
  * 20 more
  * The evidence is unclear
  * I don't know"
  (Only relevant for EmbryoGlue)
Proportion of participants with correct understanding of populations IVF add-on is applicable to | 24 hours
  "[EmbryoGlue/Intralipid/ERA test] is relevant to (tick all that apply)
  * Thin lining or thin endometrium
  * Recurrent implantation failure
  * Older female age
  * Sperm or fertilization problems
  * I don't know"
Proportion of participants with correct comprehension of cost of IVF add-on | 24 hours
  Expected cost of the add-on
  "[EmbryoGlue/Intralipid/ERA test] usually costs
  * Less than $500 AUD
  * Between $500-$1000 AUD
  * More than $1,000 AUD
  * I don't know"
Information satisfaction | 24 hours
  How satisfied participants are with the information. Items will be combined to give a composite score out of 5 (higher score = more satisfaction).
  "Please indicate below what you thought about the information for each of the below categories The information was…
  * Comprehensive
  * Important
  * Helpful
  * Trustworthy
  * Balanced
  * Clear and easy to understand" (each rated on 5-point scale from Strongly Disagree to Strongly Agree)
Emotional response | 24 hours
  Emotional response measured using the Berlin Emotional Responses to Risk instrument (Petrova 2023). Items will be combined to give a composite score out of 5 (higher score = better emotional response), with relevant items reverse scored.
  "How did you feel when you read the information about [EmbryoGlue/Intralipid/ERA test]?
  * Assured
  * Hopeful
  * Relieved
  * Anxious
  * Afraid
  * Worried" (each measured on a 5-point scale from Strongly Disagree to Strongly Agree)
  Petrova D, Cokely ET, Sobkow A, Traczyk J, Garrido D, Garcia-Retamero R. Measuring feelings about choices and risks: The Berlin Emotional Responses to Risk Instrument (BERRI). Risk Anal. 2023 Apr;43(4):724-746. doi: 10.1111/risa.13946. Epub 2022 May 23. PMID: 35606164.
Hypothetical willingness to speak to IVF specialist about using the add-on | 24 hours
  "If I was planning another IVF cycle or embryo transfer, I would speak to my IVF specialist about using [EmbryoGlue/Intralipid/ERA test]" Measured on a 5 point scale from Strongly Disagree to Strongly Agree
Self-assessed comprehension | 24 hours
  A measure of how well participant believes they understood information provided
  "After reading this information, how well do you feel you understand the potential benefits and risks of [EmbryoGlue/Intralipid/ERA test]?
  * Not at all
  * A little
  * Somewhat
  * Mostly
  * Completely"
Information length | 24 hours
  Participants perspective on whether information provided was of appropriate length "How would you rate the length of information on the website?
  * Much too short
  * A little too short
  * About right
  * A little too long
  * Much too long"
Recommend this information | 24 hours
  Whether participant would be likely to recommend the information to people considering the add-on
  "Would you recommend this information to other people having IVF who are considering [EmbryoGlue/Intralipid/ERA test]?
  * Yes
  * Maybe
  * No"

CONTACTS AND LOCATIONS:
Locations (1):
- MDHS, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
All survey data that does not contain personal data will be available
Supporting Information: Study Protocol, ICF, CSR
Time Frame: January 2026 and available for 5 years
Access Criteria: Data/information from this research project may also be used in future projects that are closely related to this project, the same general area, or could make valuable use of this data. De-identified data may be shared with other researchers upon reasonable request to Sarah Lensen.